CLINICAL TRIAL: NCT01371526
Title: Revival of Autochthonous Adrenocortical Stem Cells in Autoimmune Addison's Disease
Brief Title: Revival of Stem Cells in Addison's Study
Acronym: RoSA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Newcastle University (Other)
Responsible Party: Principal Investigator, SHS Pearce, Professor of Endocrinology, Newcastle University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RoSAv1.2:04_10: R&D#5252; 2009-018074-56 (EudraCT Number)
Record Dates: First submitted 2011-03-09; First posted 2011-06-13 (Estimated); Last update posted 2013-02-06 (Estimated); Status verified 2013-02

CONDITIONS: Adrenal Failure
MeSH Terms: conditions — Addison Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Synacthen (Experimental): active treatment
  Interventions: Drug: depot tetracosactide

INTERVENTIONS:
Drug: depot tetracosactide — 1mg, 3x weekly by sc injection

SUMMARY:
Autoimmune Addison's disease (AAD) is a rare and debilitating disease in which an autoimmune attack progressively destroys the adrenal cortex. Untreated it is universally fatal and treated people are absolutely dependent upon steroid medications lifelong, with a consequent excess in morbidity and mortality. A key feature of the adrenal cortex is that its cells are responsive to changes in circulating adrenocorticotrophic hormone (ACTH) concentration. This study aims to regenerate adrenocortical steroidogenic cell function in patients with established autoimmune Addison's disease (AAD) by stimulating proliferation and differentiation of their progenitor cells, the adrenocortical stem cells (ACSCs) (1,2). Using daily subcutaneous ACTH, administered according to two different regimens over 20 weeks, we will investigate whether regeneration of adrenal steroidogenic function through revival of ACSC activity is a realistic possibility.

ELIGIBILITY:
Inclusion Criteria:

* Established autoimmune adrenal failure for >1yr age 16 to 65

Exclusion Criteria:

* Significant cardio-respiratory, chronic renal or non-autoimmune liver disease; malignancy
* Asthma, current infectious disease, recent live vaccination, acute psychosis, peptic ulcer disease
* Pregnancy, breast feeding or plan for pregnancy within 9 months
* Known non-autoimmune cause for adrenal failure (haemorrhage, adrenoleukodystrophy etc.)
* Known hypersensitivity or allergy to Synacthen

Ages: 16 Years to 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2010-09; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Peak serum Cortisol following ACTH stimulation | Tested at 20 weeks

SECONDARY OUTCOMES:
Change in QoL | 20 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Simon H Pearce, MD, Principal Investigator — Newcastle University
Locations (1):
- Newcastle University, Newcastle upon Tyne, Tyne and Wear, United Kingdom

REFERENCES:
- [Derived] Gan EH, MacArthur K, Mitchell AL, Hughes BA, Perros P, Ball SG, James RA, Quinton R, Chen S, Furmaniak J, Arlt W, Pearce SH. Residual adrenal function in autoimmune Addison's disease: improvement after tetracosactide (ACTH1-24) treatment. J Clin Endocrinol Metab. 2014 Jan;99(1):111-8. doi: 10.1210/jc.2013-2449. Epub 2013 Dec 20. PMID 24170102